CLINICAL TRIAL: NCT02663115
Title: Influence of Severe Heart Failure to Function and Molecular Biological Parameters of Catabolism in the Human Diaphragm and Peripheral Skeletal Muscle
Acronym: LIPAMUS-HF
Status: Completed | Type: Observational
Sponsor: Norman Mangner (Other)
Responsible Party: Sponsor-Investigator, Norman Mangner, Dr. med. Norman Mangner, Heart Center Leipzig - University Hospital
Organization: Heart Center Leipzig - University Hospital (Other)
Other Study IDs: U1111-1178-1176
Record Dates: First submitted 2016-01-15; First posted 2016-01-26 (Estimated); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Heart Failure; Ischemic Myocardiopathy; Dilatative Myocardiopathy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Arm 1: Patients (age 40 - 70 years) with severe therapy-refractory heart failure caused by ischemic or dilatative myocardiopathy with indication for left ventricular assist device (LVAD) therapy
  Interventions: Other: Biopsy of the diaphragmatic muscle; Other: Skeletal muscle biopsy
- Arm 2: Patients (age 40-70 years) with the indication for elective bypass surgery and normal left ventricular function (EF>50%)
  Interventions: Other: Biopsy of the diaphragmatic muscle; Other: Skeletal muscle biopsy

INTERVENTIONS:
Other: Biopsy of the diaphragmatic muscle
Other: Skeletal muscle biopsy

SUMMARY:
Project aim is to quantify the influence of a severe therapy-refractory heart failure caused by ischemic or dilative myocardiopathy on the function of the diaphragm, its molecular biological parameters and on the M. vastus lateralis. The control group consists of patients with coronary artery disease (CAD) and normal left ventricular ejection fraction indicated for coronary artery bypass graft surgery (CABG) Differences in the geneses of heart failure (ischemic vs. dilative cardiomyopathy) will be evaluated during analysis. The ubiquitin-proteasome signaling pathway is considered as a central issue for the mechanism of the analyses muscle catabolism.

ELIGIBILITY:
Inclusion Criteria:

inclusion criteria Group A:

* age 40 - 70 years
* Restricted left ventricular pump function left ventricular ejection fraction (LVEF) > 35% on the basis of ischemic cardiomyopathy (ICM) and restricted resting cardiac output (CI> 2.4 L / min / m²)
* or restricted maximal oxygen uptake (VO2max> 17 ml / min / m²)
* Duration of heart failure> 1 year
* Maximum of individual heart failure therapy
* Heart team decision to LVAD Implantation

inclusion criteria Group B:

* age 40 - 70 years
* Restricted left ventricular pump function (LVEF) > 35% on the basis of dilatative cardiomyopathy (DCM) and restricted resting cardiac output (CI> 2.4 L / min / m²)
* or restricted maximal oxygen uptake (VO2max> 17 ml / min / m²)
* Duration of heart failure> 1 year
* Maximum of individual heart failure therapy
* Heart team decision to LVAD Implantation

inclusion criteria Group C:

* age 40 - 70 years
* coronary heart disease with indication for elective, coronary artery bypass surgery
* normal left ventricle (LV) pumping function LVEF> 50%
* stable clinical situation (no cardiac decompensation within the last 6 months)

Exclusion Criteria:

* Mechanical ventilation within the last 3 months
* Forced Expiratory Pressure (FEV1) <70% of the norm and / or therapy with α antagonists, β-mimetics or inhaled corticosteroids for the treatment of a lung disease
* Pulmonary fibrosis
* elevated diaphragm in the ultrasound or X-ray diagnosis or known paresis of the phrenic nerve
* chronic kidney disease (CKD) stage 4 and 5, i.e. glomerular filtration rate (GFR) <30ml / min / 1.73m and / or dialysis
* Acute renal failure
* Treatment with immunosuppressive agents
* Hepatic insufficiency Child-Pugh B and C
* Higher grade ventricular arrhythmias (Lown IV b)
* Acute myocardial infarction (less than three months)
* Decompensated Vitium cordis
* Age <40 years and> 70 years
* Pregnancy

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe therapy-refractory heart failure
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2016-01; Primary Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Expression of catabolic E3 ligase Muscle ring finger 1 (MuRF1) | at the time of index procedure (biopsy)

SECONDARY OUTCOMES:
in vitro measurement of the muscle protein - poly ubiquitination of Proteins | at the time of index procedure (biopsy)
in vitro measurement of the muscle protein - the proteasome activity | at the time of index procedure (biopsy)
in vitro measurement of the muscle protein - fiber typing in the muscle samples | at the time of index procedure (biopsy)
in vitro measurement of the force development of skinned muscle fibers | at the time of index procedure (biopsy)

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Center Leipzig, Leipzig, Germany

REFERENCES:
- [Derived] Mangner N, Garbade J, Heyne E, van den Berg M, Winzer EB, Hommel J, Sandri M, Jozwiak-Nozdrzykowska J, Meyer AL, Lehmann S, Schmitz C, Malfatti E, Schwarzer M, Ottenheijm CAC, Bowen TS, Linke A, Adams V. Molecular Mechanisms of Diaphragm Myopathy in Humans With Severe Heart Failure. Circ Res. 2021 Mar 19;128(6):706-719. doi: 10.1161/CIRCRESAHA.120.318060. Epub 2021 Feb 4. PMID 33535772